CLINICAL TRIAL: NCT05024435
Title: Evaluation of Semi-rigid and Flexible Catheters for Less Invasive Surfactant Administration in Preterm Infants With Respiratory Distress Syndrome - A Randomized Controlled Trial
Brief Title: Evaluation of Semi-rigid and Flexible Catheters for Less Invasive Surfactant Administration in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Lorenz Auer-Hackenberg, Medical Doctor, University Hospital Salzburg, Department of Pediatrics and Adolescent Medicine, Physician Division of Neonatology, Salzburger Landeskliniken
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 415-E/2532/7-2019
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Neonatology; Perinatal Distress Syndrome
Keywords: Less Invasive Surfactant Administration; Minimal Invasive Surfactant Treatment; Preterm Infant; Respiratory Distress Syndrome; Surfactant
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasogastric Tube (Experimental)
  Interventions: Device: Surfactant Administration
- Lisacath (Experimental)
  Interventions: Device: Surfactant Administration

INTERVENTIONS:
Device: Surfactant Administration — Laryngoscopy, intratracheal catheter placement and surfactant administration

SUMMARY:
The overall aim of this study is to determine the differences between two surfactant administration catheters in preterm infants.

DETAILED DESCRIPTION:
In this single-center, open-label, randomized-controlled trial, preterm infants requiring surfactant administration after birth, using a standardized minimal invasive protocol, were randomised to two different modes of endotracheal catheterization: Flexible Ch-4 feeding tube inserted using Magill forceps (group 1) and semi-rigid catheter (group 2). Primary outcome was duration of laryngoscopy. Secondary outcomes were complication rate and vital parameters during laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born less than 37 weeks of gestation
* Treating physician in charge of admission decides to administer intratracheal surfactant via standardized institution- LISA protocol (regardless of this study) (see Supplement file 1)
* Written informed consent signed by caregivers or legal representative to participate

Exclusion Criteria:

* Refusal to participate in study or not providing written informed consent by caregivers/parents
* Treating physician decides to use different route of surfactant administration or does not adhere to LISA protocol.
* Rupture of membranes (ROM) at less than 22 weeks of gestation or more than 6 weeks before birth
* Estimated birth weight < 3rd percentile using 2013 Fenton growth trajectories
* Twins with feto-fetal transfusion syndrome (FFTS) and FFTS being the cause of premature delivery
* Contraindications listed in the LISAcath® or Nasogastric Tube manual (esophageal/pharyngeal varices or other vascular lesions, esophageal/pharyngeal tumor, nasal fracture, skull fracture, known allergy to material)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Successful intratracheal tube Placement | Birth to 24 hours after birth

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wald, MD, Assoc. Prof., Principal Investigator — Paracelsus Medical Private University Salzburg, University Clinic of Pediatrics and Adolescent Medicine Division of Neonatology
Locations (1):
- Salzburger Landeskliniken, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Auer-Hackenberg L, Brandner J, Hofstatter E, Stroicz P, Hager T, Eichhorn A, Schutz S, Feldner R, Wald M. A pilot study of evaluation of semi-rigid and flexible catheters for less invasive surfactant administration in preterm infants with respiratory distress syndrome-a randomized controlled trial. BMC Pediatr. 2022 Nov 4;22(1):637. doi: 10.1186/s12887-022-03714-3. PMID 36333741